CLINICAL TRIAL: NCT03483064
Title: Autonomic Responses to Interferential Current in Healthy Subjects
Brief Title: Interferential Current in Lower Back
Acronym: IF-HRV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRV and interferential current
Record Dates: First submitted 2018-03-10; First posted 2018-03-29 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Lower Back
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Subjects without low back pain to whom the electric current is put but it is not activated.
- Healthy group (Experimental): Subjects without low back pain to whom the electric current is put but it is activated.
  Interventions: Other: Interferential current

INTERVENTIONS:
Other: Interferential current — interferential currents of 4,000 Hz carrier frequency, 100 Hz of AMF, for 20 minutes and with an amplitude up to the motor threshold
  Arms: Healthy group

SUMMARY:
In our daily clinical practice, one of the most frequent reasons for consultation physiotherapists is low back pain. Regardless of the origin of the problem, the approach from physiotherapy contemplates the reduction of pain through different procedures, among which all those included in electrotherapy stand out, as commented by McKenzie et al. The use of electric currents for therapeutic purposes is widespread and studied in the field of physiotherapy. However, the use of medium frequency currents, and more specifically interferential currents, provides participants with a series of important advantages, both for the patient and for the therapist.The study of low back pain in relation to treatment with interferential currents has a series of obstacles, among which the quantification of such pain and the establishment of the different parameters of the therapeutic procedure stand out. The first problem the investigators face are to objectify something that, in itself, is completely subjective: pain. In addition, pain measurement is our only guide to follow the evolution of the patient who suffers it. Another important problem, as discussed by Ward and Lucas-Toumbourou, has to do with the controversy between the different studies related to the treatment of low back pain with interferential currents.

For all the above, the approach to low back pain is complex and affects the social, labor and economic scale of the individual and society. Low back pain is the main cause of public spending for welfare and work concepts. It suffers at some point in life up to 80% of the general population and each year generates a cost equivalent to approximately between 1.7 and 2.1% of its gross domestic product in a European countries.

There is a lack of valid scientific studies on some aspects of the clinical management of low back pain and the usual clinical practice does not seem to be based strictly on the results of the researches carried out. The available data suggest that there are abuses of procedures whose benefits and risks are uncertain, while others that have proven to be more effective, safe, effective and / or efficient are underutilized. For this reason, clinical practice guidelines for non-specific low back pain have been developed in several countries in recent years. Since the first clinical practice guidelines developed in America and the United Kingdom (Quebec Task Force in 1987. In 1994, more than 30 guides who claim to be based on scientific evidence have been developed.

Electroanalgesia is a set of procedures consisting of the application of an electric current through electrodes placed on the skin of the patient in order to stimulate myelinated nerve fibers, fast driving. This activation triggers, at the central level, the implementation of descending analgesic systems of an inhibitory nature on nociceptive transmission, transported by small-caliber unmyelinated fibers. In this way, a reduction in pain is obtained. In other words, it is a question of carrying out a "differential" sensory stimulation, transcutaneously, of the tactile proprioceptive fibers, with a high speed of conduction, with the minimum response of the nociceptive fibers, of slow conduction, and of the efferent motor fibers.

The application of medium frequency interferential currents (4,000 Hz), in addition to reducing the pain caused by the stimulation of thick nerve fibers, produces the normalization of the neurovegetative balance. According to De Domenico, this means a cushioning of the orthosympathetic system, which is reflected in muscle relaxation and improved circulation, which also helps to reduce pain.

But the clinical impact of interferential currents on non-specific chronic low back pain remains poorly studied. Thus, clinical trials show some controversy and support its efficacy in combination with other treatments. A systematic review found that the interferential current demonstrates advantages over placebo and without treatment when associated with exercises and massages. In contrast, the European clinical practice guideline for the treatment of chronic low back pain concluded that there was no evidence of its effectiveness compared to sham intervention or placebo. However, recent studies of a randomized clinical trial with interferential currents on patients with nonspecific chronic low back pain report very favorable results in terms of the reduction of perceived pain and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* subjects without low back pain
* Not being doing another type of physical therapy.

Exclusion Criteria:

* Presence of neurological, musculoskeletal or sensory disorder.
* Infectious, febrile or hypotensive processes.
* Appreciation to the application of electrotherapy, measured through the EAPP scale

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Hear rate variability | 1 day
  NN interval series, measured by sympathetic-parasympathetic balance

CONTACTS AND LOCATIONS:
Locations (1):
- Blanca de La Cruz Torres, Seville, Spain

REFERENCES:
- [Derived] De-la-Cruz-Torres B, Martinez-Jimenez E, Navarro-Flores E, Palomo-Lopez P, Abuin-Porras V, Diaz-Meco-Conde R, Lopez-Lopez D, Romero-Morales C. Heart Rate Variability Monitoring during Interferential Current Application in the Lower Back Area: A Cross-Sectional Study. Int J Environ Res Public Health. 2021 Mar 25;18(7):3394. doi: 10.3390/ijerph18073394. PMID 33805948